CLINICAL TRIAL: NCT06470854
Title: Nebulized Dexmedetomidine for Post-dural Puncture Headache: A Comparative Case-Control Study Versus Bilateral Greater Occipital Nerve Block
Brief Title: Effect of Nebulized Dexmedetomidine on Post-dural Puncture Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Lotfy, Assistant Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR665/4/24
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group One (Active Comparator)
  Interventions: Drug: Nebulized Dexmedetomidine
- Group Two (Active Comparator)
  Interventions: Procedure: Bilateral greater occipital nerve block

INTERVENTIONS:
Drug: Nebulized Dexmedetomidine — Nebulized Dexmedetomidine was prepared to provide 1 µg/kg and the calculated dose of DXM was diluted by 4-ml of 0.9% saline and was provided in the nebulizer to be nebulized in twice daily; i.e. every 12 hours for 72 hours
  Arms: Group One
Procedure: Bilateral greater occipital nerve block — The injection solution was prepared by mixing 2-ml of 2% lidocaine with 2-ml (8 mg) of dexamethasone. A line was drawn extending between the mastoid process and the external occipital protuberance, this line was divided as a medial third and lateral two-thirds to localize the occipital artery and the greater occipital nerve was located on the medial side of the artery where it exits out of the trapezius fascia into the nuchal line about 5-cm lateral to midline and injection was performed bilaterally to achieve bilateral block.
  Arms: Group Two

SUMMARY:
Dural puncture during neuroaxial procedures is the most frequent major complication that causes the development of post-dural puncture headache (PDPH) in 16%-86% of cases. PDPH could be defined as severe positional headache that usually presents during the first 72-h following accidental dural puncture.

Dexmedetomidine (DXM) is a potent and highly selective α2-adrenergic agonist that was approved for ICU and procedural sedation in adults. Additionally, DXM has pleiotropic effects for its sympatholytic, amnestic, and analgesic properties. Regarding routes of administrations, DXM allows high flexibility and can be administered through intravenous (IV), intramuscular, buccal, intranasal and inhalational routes.

Nebulized DXM at 1 µg/kg is a favorable alternative to the intravenous route in short duration surgeries because it attenuates heart rate response to laryngoscopy. However, the effects of nebulized DXM on blood pressure are controversial.

it was assured that it has a role in reduction of the intraoperative anesthetic requirements and analgesic consumption.

The prophylactic and management strategies for PDPH are heterogeneous because of the absence of clear guidelines and protocols for the management of PDPH. However, the general plan for PDPH management consists of conservative treatment and if failed invasive procedures such as blood patch were applied.

ELIGIBILITY:
Inclusion Criteria:

* Women had CS under spinal anesthesia;
* Women started to complain of PDPH;
* Women were free of exclusion criteria.

Exclusion Criteria:

* Women had prior history of PDPH or headache for any cause;
* Women had essential hypertension;
* Women with previous history of habitual hypotension or accidental syncope secondary to postural hypotension;
* Women with tempromandibular disorders;
* Women who refused to participate in the study were excluded.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
The extent of reduction of consumed analgesia | 5 Months
  Efficacy of both modalities for relieve of Post Dural Puncture Headache in the women who included in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El Gharbyia, Egypt